CLINICAL TRIAL: NCT04592302
Title: The Impact of Smoking on Outcomes and Complications in Total Joint Arthroplasty: A Prospective Crossover Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: LAUS16D.265
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Smoking; Total Joint Arthroplasty
MeSH Terms: conditions — Smoking | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking Cessation Group: participants are required to cease smoking for 4 weeks prior to and 2 weeks after TJA without any nicotine replacement (any other smoking cessation aids the patient chooses will be allowed)
  Interventions: Diagnostic Test: Blood Draw
- Smoker Group 2: participants who are allowed to continue smoking and using nicotine in any form at their own discretion during the perioperative period
  Interventions: Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: Blood Draw — 2-4 weeks before surgery a blood draw will be taken to test for nicotine levels in the body

SUMMARY:
The purpose of this study is to examine the impact of smoking cessation on total joint arthroplasty patients with respect to perioperative complications and outcomes. The investigators will examine patients who are asked to stop smoking in any manner they choose and also refrain from nicotine replacement therapy, and those who are allowed to continue smoking during the perioperative period for their total knee or total hip replacement.

ELIGIBILITY:
Inclusion criteria:

1. Primary elective total joint arthroplasty patients undergoing surgery with a Rothman Institute arthroplasty surgeon.
2. Participant is a current smoker.
3. Diagnosis of osteoarthritis, inflammatory arthritis, and post-traumatic arthritis.

Exclusions criteria:

1. Age < 18
2. Revision surgery
3. Prior infection in hip or knee at the surgical site
4. BMI >40 (It is currently the standard of care in our practice to require patients to have a BMI < 40 due to an increased risk of infection. This will not represent a change in practice.)
5. Diabetics with Hgb A1C >8 (It is currently the standard of care in our practice to require patients to have a Hgb A1C <8 due to an increased risk of infection. This will not represent a change in practice.)
6. Patients using chewing tobacco, cigars, or other form of oral tobacco product
7. Patients using e-cigarettes or vaporizers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are current smokers having surgery for total joint arthroplasty at Rothman Orthopaedic Institute
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 3 months
  The primary objective of this study is to examine the impact of smoking cessation on total joint arthroplasty patients with respect to combined complications. For the purpose of the study combined complications will include: major in-hospital complications (MI, CVA, PE, pneumonia, return to the operating room, mortality), wound complications, readmission at 90 days, 90-day major complications (MI, CVA, PE, pneumonia, return to the operating room, mortality), and wound complications (prolonged hospitalization due to a wound issue, prolonged drainage > 7 days, superficial or deep SSI

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States